CLINICAL TRIAL: NCT03235323
Title: Study of Efficacy of External CounterPulsation on Reducing the Prevalence of Vein Graft Failure and Improving Cardiac Function for Postoperative Coronary Artery Bypass Grafting Patients
Brief Title: Efficacy of External CounterPulsation for Postoperative Coronary Artery Bypass Grafting Patients
Acronym: SEECABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mengya Liang (Other)
Responsible Party: Sponsor-Investigator, Mengya Liang, Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LS2017-144
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Counterpulsation; Coronary Artery Bypass
Keywords: Vein Graft Failure; Coronary Artery Bypass; External Counterpulsation
MeSH Terms: interventions — Counterpulsation

STUDY DESIGN:
Intervention Model Description: A standard ECP protocol involves 35 one-hour sessions (once per day, 5 days a week) and continuous for 7 weeks. ECP consists of three sets of pneumatic cuffs attached to each of the patient's legs at the calf and lower and upper thigh. The inflation of the cuffs is triggered by a computer, and timing of the inflation is based on the R wave of the electrocardiogram. The ECP therapist adjusts the inflation and deflation timing to provide optimal blood movement per a finger plethysmogram waveform reading.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECP group (Experimental): Patients of ECP group are subjected to a standard ECP protocol one week postoperatively. A standard ECP protocol involves 35 one-hour sessions (once per day, 5 days a week) and continuous for 7 weeks. ECP consists of three sets of pneumatic cuffs attached to each of the patient's legs at the calf and lower and upper thigh. The inflation of the cuffs is triggered by a computer, and timing of the inflation is based on the R wave of the electrocardiogram. The ECP therapist adjusts the inflation and deflation timing to provide optimal blood movement per a finger plethysmogram waveform reading.
  Interventions: Device: External Counterpulsation
- Control group (No Intervention): Patients of Control group received routine medicine treatment postoperatively

INTERVENTIONS:
Device: External Counterpulsation — ECP is a non-invasive method which consists of three sets of pneumatic cuffs attached to each of the patient's legs at the calf and lower and upper thigh. The inflation of the cuffs is triggered by a computer, and timing of the inflation is based on the R wave of the electrocardiogram. The ECP therapist adjusts the inflation and deflation timing to provide optimal blood movement per a finger plethysmogram waveform reading. This produces a retrograde flow of blood in the aorta resulting in a diastolic augmentation of blood flow and also an increase in venous return, which leads to an improved coronary perfusion pressure during diastole.
  Arms: ECP group

SUMMARY:
The aim of this study is to evaluate the effect of External CounterPulsation on postoperative heart function and vein graft failure rates of coronary artery bypass grafting patients.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is prevalent worldwide and the leading cause of mortality of citizens. Coronary Artery Bypass Grafting (CABG)is one of the major revascularization procedures for multi-vessel disease nowadays. However vein graft failures (VGF) are known to occur frequently following CABG surgery . It is estimated that VGF developed in 25% patients in half a year postoperatively, and up to 50% vein grafts would result in occlusion in ten years postoperatively. Surgical success depends on the continued patency of grafts, and VGF has been associated with worse outcomes in CABG patients. Thus prevention of VGF following CABG is an active area of scientific inquiry. External counter pulsation (ECP) is a non-invasive method which consists of three sets of pneumatic cuffs attached to each of the patient's legs at the calf and lower and upper thigh. The inflation of the cuffs is triggered by a computer, and timing of the inflation is based on the R wave of the electrocardiogram. The ECP therapist adjusts the inflation and deflation timing to provide optimal blood movement per a finger plethysmogram waveform reading. This produces a retrograde flow of blood in the aorta resulting in a diastolic augmentation of blood flow and also an increase in venous return, which leads to an improved coronary perfusion pressure during diastole.ECP has been elucidated that it may release angina symptoms and improve the prognosis of CAD, however, it remained unknown that weather EECP can reduce VGF rates following CABG surgery. The aim of this study is to evaluate the effect of ECP on heart function of CABG patients and VGF rates.

To address this investigation, patients underwent CABG with at least one vein graft are enrolled and randomize them into control or ECP group, the ECP intervention will be carried out with a standard protocol which involves 35 one-hour sessions (5 days a week) for continuous 7 weeks, and the follow-up will last for 2 years. The primary endpoints are the 2-year major composite cardiovascular events (MACEs,) and 2-year vein graft patency rate determined by coronary CT angiography, secondary endpoints include scoring of angina pectoris, heart function by echocardiography, biomarkers of arteriosclerosis and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent coronary artery bypass grafting surgery

Exclusion Criteria:

* Cerebral hemorrhage within six months;
* Obvious aortic insufficiency;
* Aortic aneurysm;
* Aortic dissection;
* Coronary fistula or severe coronary aneurysm;
* Symptomatic Congestive heart failure
* New York Heart Association（NYHA）heart function class IV
* Valvular heart disease;
* Congenital heart diseases;
* Cardiomyopathies
* Uncontrolled hypertension, defined as SBP≥180mmHg or DBP≥110mmHg;
* Lower limb infection;
* Deep venous thrombosis;
* Progressive malignancies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-08-07 (Estimated); Study Completion 2021-08-07 (Estimated)

PRIMARY OUTCOMES:
2-year vein graft patency rate | Two years postoperatively
  2-year vein graft patency rate determined by coronary CT angiography
2-year major composite cardiovascular events (MACEs) | Two years postoperatively
  2-year major composite cardiovascular events,including STEMI/NSTEMI，readmission of heart attack, renal dialysis and acute heart failure

SECONDARY OUTCOMES:
Canadian Cardiovascular Society （CCS） scoring | One and two years postoperatively
left ventricular end-systolic volume index (LVESVI) and Ejection Fraction | One and two years postoperatively
  left ventricular end-systolic volume index (LVESVI) and Ejection Fraction by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Zhongkai Wu, Study Director — Department of Cardiovascular Medcine
Locations (1):
- Department of cardiac surgery, The first affiliated hospital of Sun Yat-sen university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang Y, He X, Chen X, Ma H, Liu D, Luo J, Du Z, Jin Y, Xiong Y, He J, Fang D, Wang K, Lawson WE, Hui JC, Zheng Z, Wu G. Enhanced external counterpulsation inhibits intimal hyperplasia by modifying shear stress responsive gene expression in hypercholesterolemic pigs. Circulation. 2007 Jul 31;116(5):526-34. doi: 10.1161/CIRCULATIONAHA.106.647248. Epub 2007 Jul 9. PMID 17620513